CLINICAL TRIAL: NCT06701253
Title: Ultrasound of the Anterior Neck Tissues, as a New Tool in the Evaluation of Difficult Airway.
Brief Title: Upper Airway Ultrasound Evaluation
Status: Recruiting | Type: Observational
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Agathi Karakosta, Assistant Professor of Anaesthesiology, University of Ioannina
Other Study IDs: 768
Record Dates: First submitted 2024-11-03; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Airway Management; Point of Care; Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: point of care ultrasound — Point of care ultrasound for upper airway evaluation.

SUMMARY:
Current guidelines support the use of predictive clinical tests in the evaluation of difficult airway, meaning either difficult bag and mask ventilation, conventional laryngoscopy and/or endotracheal intubation. However, despite the clinical use of these predictive tests, unpredictive difficult laryngoscopy complicates 1.5-13% of cases. Life threatening scenarios may be encountered in patients with difficult or impossible bag and mask ventilation.

Anaesthesiologists are familiar with the use of ultrasound, with peripheral nerve blockade and central vascular access representing the most popular applications during the last decades. The ultrasound provides real time and accurate images. According to the current literature, there are only a handful of studies relevant to the application of point of care ultrasound (POCUS), as a new tool in the upper airway evaluation. It is a new field of research with high interest.

This is a prospective observational study to investigate if specific ultrasound measurements of the anterior neck can serve as predictors of difficult airway. The ultrasound parameters will be measured preoperatively, during the preanaesthetic evaluation, along with standard clinical prognostic tools, like the mallampati score. The ultrasound parameters to be investigated are:

1. the distance from thyroid isthmus to skin surface,
2. the distance from the hyoid bone to the skin surface,
3. the distance from the anterior commissure of vocal cords to the skin surface,
4. the distance from skin to the trachea at the level of jugular notch,
5. the distance from skin to epiglottis corresponding to half of the distance between thyroid cartilage and hyoid bone,
6. and the angle between glottis and epiglottis. After the induction in anaesthesia, the Cormack Lehane score (grading of the laryngoscopy view) and the Han scale (grading of the degree of difficulty of bag and mask ventilation) will also be recorded.

The goal of this study is the investigation of the role of POCUS in the evaluation of difficult bag and mask ventilation and difficult intubation. The primary endpoint is the incidence of difficult bag and mask ventilation and the incidence of difficult laryngoscopy and intubation. Secondary endpoints are the correlations between clinical prognostic tools of difficult airway and the POCUS parameters under investigation.

DETAILED DESCRIPTION:
Ultrasound of the anterior neck tissues, as a new tool in the evaluation of difficult airway.

Introduction The current guidelines provide predictive clinical tests in the evaluation of difficult airway, relevant to the mask ventilation, conventional laryngoscopy and endotracheal intubation. Despite similarities in predictors, the incidence of mask ventilation is distinct from difficult laryngoscopy and intubation, 7.8% and 12.3% respectively.

However, despite the clinical use of these predictive tests, unpredictive difficult laryngoscopy complicates 1.5-13% of cases. The risk of life-threatening complications is increased in patients with difficult or impossible bag and mask ventilation.

Anaesthesiologists are familiar with the use of ultrasound, with peripheral nerve blockade and central vascular access representing the most popular applications of the last decades. Ultrasound provides quick, easy and accurate images.

According to the current literature, there are a few studies relevant to the application of point of care ultrasound (POCUS), as a new tool in the upper airway evaluation. It is a new field of research with high interest.

This is a prospective observational study which is taking place at the University Hospital of Ioannina in order to investigate if some ultrasound measurements of the anterior neck can serve as predictors of difficult airway. The goal is to investigate the role of POCUS in the evaluation of difficult bag and mask ventilation and difficult intubation.

Aim of the study The primary outcome of this study is the incidence of difficult bag and mask ventilation and the incidence of difficult laryngoscopy and intubation.

Difficult bag and mask ventilation is defined as the inability of an unassisted conventionally trained anesthesiologist to maintain the oxygen saturation as measured by pulse oximetry > 92% or to prevent or reverse signs of inadequate ventilation during positive-pressure mask ventilation under general anesthesia.

Difficult intubation is when a conventionally trained anesthesiologist needs more than 3 attempts or more than 10 min to intubate the patient.

Secondary outcome is the investigation of the relationship between ultrasound parameters, Cormack- Lehane scale, Han scale and the clinical prognostic tools.

Secondary endpoints are the investigations of the relationships between standard clinical prognostic tools of difficult airway and the POCUS parameters under investigation.

Materials and Methods Anesthetic technique The ultrasound parameters will be measured in all the participants in the preanesthetic evaluation. The rest of anesthetic management will follow the standard practices and the protocols of our Anaesthesiology Department.

Data collection The collection of data concerns two time periods. The first, during the preanesthetic evaluation, when the standard clinical prognostic markers of difficult airway (Mallampati score, thyromental distance, sternomental distance, mouth opening, neck circumference, upper lip bite test, cervical mobility, presence of beard), as well as somatometrics (age, weight, height, gender and race) will be recorded. Moreover, the type of the operation, the physical classification of the American Society of Anesthesiologists physical status (ASA score) score, the comorbidities (by application of the Charlson Comorbidity Index) and the history of Obstructive Sleep Apnea (as evaluated by the Stop-Bang questionnaire) will also be recorded preoperatively.

Lastly, specific ultrasound markers of the anterior neck tissue will be evaluated preoperatively. This investigation will include the recognition and measurement of the following ultrasound parameters, either with the probe in the transverse or the sagittal axis:

1. the distance from thyroid isthmus to skin surface (transverse axis),
2. the distance from the hyoid bone to the skin surface (transverse axis),
3. the distance from the anterior commissure of vocal cords to the skin surface (transverse axis),
4. the distance from skin to the trachea at the level of jugular notch (transverse axis)
5. the distance from skin to epiglottis corresponding to half of the distance between thyroid cartilage and hyoid bone (sagittal axis),
6. and the angle between glottis and epiglottis (sagittal axis). The second period of data collection involves the post induction of general anaesthesia and intubation period. At this point the Cormack-Lehane score (grading of the laryngoscopy view), the Han scale (grading of the degree of difficulty of bag and mask ventilation), the total number of intubation attempts with conventional laryngoscopy, the number of the anesthesiologists involved and their level of experience, the use of auxiliary tools (McCoy laryngoscope, ESCHMANN bougie, forceps Magille, supraglottic devises, video laryngoscope, and other relevant tools), the kind and the size of the endotracheal tube and the outcome (successful conventional endotracheal intubation, postponing operation, front of neck access, etc.) will be recorded in detail.

Size sample and statistical analysis This is a prospective observational study. The sample size is calculated by the incidence of difficult intubation and laryngoscopy according to current literature. Specifically, the incidence of difficult intubation in the operation theatre varies between 1.15 up to 3.8% and the incidence of difficult laryngoscopy between 6.1 up to 13%.

Our aim is to include 60 cases in our study (10 per ultrasound parameter) with difficult intubation/laryngoscopy. To achieve this goal, we need to include 460 to 980 cases, based on the above-mentioned minimum and maximum reported incidences of difficult laryngoscopy. However, recruitment will be completed when at least 60 cases of difficult laryngoscopy and/or difficult intubation have been recorded.

The data analysis will be performed using the software Stata tm (Version 10.1 MP, Stata Corporation, College Station, TX 77845, USA).

ELIGIBILITY:
Inclusion Criteria: age>18, elective surgery under general anesthesia with endotracheal intubation

Exclusion Criteria:

* obstetric surgeries,
* pregnancy,
* non elective surgeries,
* patients with previous surgeries involving the anterior surface of the neck (i.e., thyroid surgery),
* patients with history of cervical radiation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General surgical population.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-11-18 (Estimated); Study Completion 2025-06-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of difficult intubation | From the beginning of the pre-oxygenation period up to securing the airway, with either up to 3 attempts of conventional laryngoscopy/intubation, or non-conventional intubation, or waking up the patient, whichever comes first.
  Difficult intubation is defined as requirement of more than three attempts with conventional laryngoscopy.
Incidence of difficult bag and mask ventilation | From the beginning of the pre-oxygenation period up to securing the airway, with either up to 3 attempts of conventional laryngoscopy/intubation, or non-conventional intubation, or waking up the patient, whichever comes first.
  Difficult mask ventilation is defined as the inability of an unassisted anesthesiologist to maintain the measured oxygen saturation as measured by pulse oximetry > 92% or to prevent or reverse signs of inadequate ventilation during positive-pressure mask ventilation under general anesthesia.

SECONDARY OUTCOMES:
Cormack-Lehane classification | From the beginning of the pre-oxygenation period up to the first, second or third attempt of conventional laryngoscopy, whichever comes first.
  Classifies laryngoscopy views obtained by direct laryngoscopy based on the structures seen (Grade I: visualization of the entire laryngeal aperture; Grade II: visualization of only the posterior commissure of the laryngeal aperture; Grade III: visualization of only the epiglottis; Grade IV: visualization of only the soft palate).
Han scale classification | From the beginning of the pre-oxygenation period up to securing the airway, with either up to 3 attempts of conventional laryngoscopy/intubation, or non-conventional intubation, or waking up the patient, whichever comes first.
  Classifies the difficulty in bag and mask ventilation (Grade I: easy mask ventilation, Grade II: needs oral airway or adjuvant with or without neuromuscular blocking agents, Grade III: difficult - inadequate or unstable or requiring two care providers, with or without neuromuscular blocking agents, Grade IV: impossible - unable to mask ventilate with or without neuromuscular blocking agents).
Distance from thyroid isthmus to skin surface | 24 hours before elective surgery and general anaesthesia needing endotracheal intubation, during the pre-anesthetic visit.
  Ultrasound measurement of the distance from thyroid isthmus to skin surface with the probe in the transverse axis.
Distance from hyoid bone to skin surface | 24 hours before elective surgery and general anaesthesia needing endotracheal intubation, during the pre-anesthetic visit.
  Ultrasound measurement of the distance from hyoid bone to skin surface with the probe in the transverse axis.
Distance from anterior commissure to skin surface | 24 hours before elective surgery and general anaesthesia needing endotracheal intubation, during the pre-anesthetic visit.
  Ultrasound measurement of the distance from anterior commissure of vocal cords to the skin surface with the probe in the transverse axis.
Distance from trachea to skin surface | 24 hours before elective surgery and general anaesthesia needing endotracheal intubation, during the pre-anesthetic visit.
  Ultrasound measurement of the distance from trachea to skin surface at the level of jugular notch with the probe in the transverse axis.
Distance from epiglottis to skin surface | 24 hours before elective surgery and general anaesthesia needing endotracheal intubation, during the pre-anesthetic visit.
  Ultrasound measurement of the distance from epigottis to skin at the level of the thyrohyoid membrane with the probe in the sagital axis.
Angle between the epiglottis and glottis | 24 hours before elective surgery and general anaesthesia needing endotracheal intubation, during the pre-anesthetic visit.
  Ultrasound measurement of the angle between epiglottis and glottis at the level of thyrohyoid membrane with the probe in the sagital axis.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Ioannina, Ioannina, Epirus, Greece

IPD SHARING:
Plan to Share IPD: Undecided